CLINICAL TRIAL: NCT02566252
Title: A Randomized, Open-label, Crossover Study to Assess the Safety, Tolerability, and Pharmacodynamics of PUL-042 Inhalation Solution in Healthy Subjects and the Effect of Pretreatment With Cromolyn Sodium or Albuterol Sulfate
Brief Title: Effect of Pre-Treatment With Cromolyn or Albuterol on Response to PUL-042 Inhalation Solution (PUL-042)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pulmotect, Inc. (Industry)
Collaborators: WCCT Global (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PUL-042-003
Record Dates: First submitted 2015-09-29; First posted 2015-10-02 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Healthy
Keywords: Safety; tolerability
MeSH Terms: interventions — Cromolyn Sodium; Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PUL-042 (Experimental): PUL-042 Inhalation Solution
  Interventions: Drug: PUL-042 Inhalation Solution
- Cromolyn sodium (Experimental): Pre-Treatment with cromolyn sodium followed by PUL-042 Inhalation Solution Administration
  Interventions: Drug: PUL-042 Inhalation Solution; Drug: Cromolyn Sodium
- Albuterol sulfate (Experimental): Pre-Treatment with albuterol sulfate followed by PUL-042 Inhalation Solution Administration
  Interventions: Drug: PUL-042 Inhalation Solution; Drug: Albuterol sulfate

INTERVENTIONS:
Drug: PUL-042 Inhalation Solution — PUL-042
Drug: Cromolyn Sodium — Pre-treatment
  Arms: Cromolyn sodium
Drug: Albuterol sulfate — Pre-treatment
  Arms: Albuterol sulfate

SUMMARY:
This study evaluates the effect of pre-treatment with either cromolyn sodium or albuterol sulfate on the safety and tolerability or PUL-042 Inhalation Solution in healthy subjects.

DETAILED DESCRIPTION:
Healthy subjects (8 per cohort) will be randomized to either pre-treatment or no pre-treatment (4 per group). The initial cohort will receive pre-treatment with cromolyn sodium. Subjects will be followed for 2 weeks for safety and tolerability, undergo a 2 week washout period and then be assigned to the alternative treatment (i.e., subjects who received cromolyn sodium prior to PUL-042 inhalation solution will not receive pretreatment) and then followed for an additional 2 weeks.

Subsequent cohort will receive pre-treatment with albuterol sulfate in a like manner.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of non-childbearing potential (defined as surgically sterilized [tubal ligation/hysterectomy/bilateral salpingo oophorectomy or post- menopausal for > 2 years) with a negative urine human chorionic gonadotropin (hCG) pregnancy test at the Screening Visit
* Body Mass Index (BMI) between 18 and 30 kg/m2
* Ability to perform spirometry according to American Thoracic Society standards
* Normal spirometry (forced expiratory volume in 1 second [FEV1] and forced vital capacity [FVC] ≥ 80% and ≤ 120% based on predicted values) at the Screening Visit and at Visit 2.
* Pulse oximetry ≥95% on room air
* Ability to understand and give informed consent
* Males willing to practice contraception (condom + spermicide) during the study and for 30 days after completion of the

Exclusion Criteria:

* Febrile (temperature ≥ 99.5°Fahrenheit)
* A history of use of any tobacco products during the year prior to the Screening Visit and a total exposure of > 5 pack years or a positive urine cotinine level at the Screening Visit
* Clinically significant laboratory finding as determined by the Principal Investigator or designee at the Screening Visit or at Visit 2
* Positive test for drugs of abuse (alcohol, cannabinoids, opiates, cocaine, amphetamine, barbiturates, benzodiazepine, phencyclidine)
* Any active medical problems requiring treatment
* Subjects who exhibit symptoms of respiratory infection or have experienced respiratory symptoms of an upper respiratory infection within 30 days prior to the Screening Visit.
* History of chronic pulmonary disease (eg, asthma [including atopic asthma, exercise induced asthma, or asthma triggered by respiratory infection], pulmonary fibrosis), pulmonary hypertension, or heart failure
* Any out of range QTc Fridericia (QTcF) or other clinically significant ECG findings as determined by the Principal Investigator or designee at Visit 2 or Visit 12.
* History of atopic reactions
* Administration of any anti-inflammatory therapy (eg, no steroidal anti-inflammatory drugs or corticosteroids) within 4 weeks prior to randomization or expected to be ongoing during the study
* An anticipated need for use of any inhaled medication during the study
* Intake of coffee, tea, cola drinks, chocolate on days of Study Visits 1-21
* Intake of alcohol, caffeine or strenuous exercise within 72 hours prior to study drug administration or intake of grapefruit within 7 days prior to the administration of study drug
* Intake of alcohol within 4 hours of spirometry; smoking within 1 hour of spirometry; performing vigorous exercise within 30 minutes of spirometry; wearing clothing that substantially restricts full chest and abdominal expansion; or eating a large meal within 2 hours of spirometry
* Administration of any over the counter (OTC)/prescription medication, supplements, herbals or vitamins within 14 days prior to study drug administration. Administration of Tylenol within 72 hours of study drug administration (doses up to 2g/day will be allowed prior to 72 hours before study drug administration)
* Exposure to any investigational agent within 30 days prior to the Screening Visit
* Receipt of a flu vaccine in the last 3 months
* Prior exposure to PUL-042
* Known positive for human immunodeficiency virus, or on active anti-retroviral therapy and known hepatitis B surface antigen positive or hepatitis C positive

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent, treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE v4.0) | 6 weeks

OTHER OUTCOMES:
Effect of pre-treatment with cromolyn sodium or albuterol sulfate on serial forced expiratory volume in 1 second (FEV1) from 0-8 hours post PUL-042 administration | 8 hours
  Area under the FEV1 curve from dosing until 8 hours post-dose (AUC0-8)
Number of participants with FEV1 decrease of > 12% compared to pred-dose baseline | 2 weeks
  Serial measurements of FEV1
Number of participants with absolute neutrophil count (ANC) outside the normal range | 2 weeks
  Serial measurements of ANC

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Ababa, MD, Principal Investigator — West Coast Clinical Trials
Locations (1):
- WCCT Global, Cypress, California, United States